CLINICAL TRIAL: NCT01210235
Title: FLU-FIT Program at Kaiser Permanente Northern California
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RSGPB-09-010-01-CPPB
Record Dates: First submitted 2010-09-25; First posted 2010-09-28 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer screening; preventive health; primary care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLU-FIT Arm (Experimental): In this arm, eligible patients aged 50-75 will be offered a FIT kit
  Interventions: Behavioral: FLU-FIT Program
- FLU-Only Arm (No Intervention): In this arm, patients will receive flu shots as usual, without the FLU-FIT intervention.

INTERVENTIONS:
Behavioral: FLU-FIT Program — In the intervention, eligible patients aged 50-75 who come in for flu shots and are due for colorectal cancer screening will be offered FIT.
  Arms: FLU-FIT Arm

SUMMARY:
The investigators overall goal is to develop, implement, test, and disseminate an intervention to increase colorectal cancer screening rates at Kaiser Permanente (KP) by providing home fecal immunochemical test kits (FIT) to eligible patients aged 50 and older who participate in annual influenza vaccination campaigns. The investigators hypothesis is that the FLU-FIT Program will be an effective method to increase colorectal cancer screening rates at Kaiser Permanente.

DETAILED DESCRIPTION:
Background: Colorectal cancer is the second leading cause of cancer death in the U.S. Many of these deaths could be prevented by screening, which is recommended for adults aged 50 and older. Effective screening options include yearly fecal occult blood tests, flexible sigmoidoscopy every 5 years, or colonoscopy every 10 years. Unfortunately, despite these recommendations and options, only half of adults aged 50 and older are up to date with any test. Simple, cost-effective approaches to increase colorectal cancer screening rates are needed to reduce the burden of colorectal cancer in the U.S.

Objective/Hypothesis: Our hypothesis is that offering annual colorectal cancer screening with fecal occult blood tests to eligible adults aged 50 and over during annual nurse-run influenza vaccination clinics will result in increased colorectal cancer screening rates, reaching populations that have been under-screened in the past. Our overall objective is to develop, implement, test, and disseminate this intervention using an annual fecal immunochemical test for occult blood (FIT) at Kaiser Permanente (KP) Northern California.

Specific Aims: The specific aims of this research are to (1) develop and implement a comprehensive nurse-run FLU-FIT Program at the KP Santa Clara facility that will systematize the offering of FIT to all eligible patients aged 50 to 80 who attend annual influenza vaccination clinics; (2) test the effectiveness of the FLU-FIT Program in improving colorectal cancer screening rates in the context of a time-randomized, controlled trial involving an ethnically diverse population of influenza vaccination clinic attendees at 8 influenza vaccination sites within 4 other KP Northern California service areas; (3) evaluate the reach and robustness of the FLU-FIT Program as implemented within these 8 sites, and (4) create a FLU-FIT Program Toolkit that can be used in further efforts to disseminate this intervention both within Kaiser Permanente and to other clinical settings.

Study Design: The study will be conducted in 3 phases. In Phase 1 (Year 1), we will evaluate a pilot FLU-FIT Program that is already underway at KP Santa Clara and implement it systematically for its annual influenza vaccination clinics in 2009-2010. In Phase 2 (Years 2 and 3), the key elements of the KP Santa Clara FLU-FIT Program will be tested in a time-randomized trial within 8 other KP Northern California sites. On randomly assigned dates at each of the 8 influenza vaccination clinic sites, patients will receive either the FLU-FIT Program (intervention) or influenza vaccination only (control). The primary outcome will be the proportion of intervention subjects between the ages of 50 and 80 who are initially due for colorectal cancer screening that become up to date with colorectal screening within 3 months after receiving their influenza vaccine, as compared to similar subjects in the control group. The robustness of the intervention as an effective and sustainable intervention to increase rates of colorectal cancer screening in "real world" settings will also be evaluated according to the RE-AIM criteria (Reach, Efficacy, Adoption, Implementation, and Maintenance). In Phase 3 (Year 4), data will be analyzed, and a toolkit for further dissemination activities will be developed.

Cancer Relevance: If successful and widely implemented, the FLU-FIT Program could increase access to colorectal cancer screening for millions of Americans. This approach could also provide a model for developing effective cancer screening interventions that do not depend solely on the primary care clinician, and that can be triggered by other regular contacts that patients have with the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50-75 at the time of their flu shots who are also due for colorectal cancer screening.

Exclusion Criteria: none

-

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7465 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Completion of colorectal cancer screening by eligible patients within 3 months of their flu shot | from time of getting flu shot until 3 months later
  We will determine the proportion of patients aged 50-75 who are eligible for colorectal cancer screening at the time of their annual flu shot and become up to date with colorectal cancer screening 3 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Potter, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States